CLINICAL TRIAL: NCT01392144
Title: Phase II Evaluation of Exhaled Nitric Oxide as a Predictive Biomarker for Radiation Pneumonitis
Brief Title: Phase II Evaluation of Exhaled Nitric Oxide (NO)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2010-0446; R21CA159105 (Other: NIH)
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: Radiation pneumonitis; RP; Nitric oxide; NO; Thoracic; Esophagus cancer; Lung cancer; Radiation therapy; radiotherapy; RT; XRT; Airway; Alveolar; Nitric oxide breath analyzer; Questionnaires
MeSH Terms: conditions — Lung Neoplasms; Radiation Pneumonitis; Esophageal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nitric Oxide Breath Analysis: Nitric Oxide Breath Test + Questionnaires
  Interventions: Procedure: Nitric oxide breath test; Behavioral: Questionnaires

INTERVENTIONS:
Procedure: Nitric oxide breath test — Breathe out into a device (nitric oxide breath analyzer) for 10 seconds; repeated 3 times. Done prior to start of radiation therapy, 1 week before completion of radiation therapy, at completion of radiation therapy, then at each follow-up visit for 6 months.
Behavioral: Questionnaires — On day of each breathing test, completion of a breathing and symptom questionnaire, approximately 10 minutes.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if the level of nitric oxide you breathe out may relate to the amount of breathing complications that you may experience due to radiation treatment.

DETAILED DESCRIPTION:
Nitric Oxide Breathing Test:

If you agree to take part in this study, you will have a nitric oxide breathing test performed before, during and after radiation therapy. You will you will have a nitric oxide breathing test 1 week before you complete radiation therapy, when you complete radiation therapy, and at each follow-up visit for 6 months.

To complete this test, you will breathe out into a device called a nitric oxide breath analyzer for 10 seconds. You will repeat this test 3 times. The results of this test will give researchers information about possible inflammation in your lungs. The results of this test will be compared with any breathing symptoms you may experience during the same time period.

For your first breath testing session and any session when your nitric oxide level is at least 1 ½ times higher than the first session, you will repeat the test for up to 5 different "breathe out rates". This additional testing will allow the researchers to find where in your lungs the nitric oxide increase is coming from.

Breathing Symptoms Questionnaire:

On the day of each breathing test, you will complete a questionnaire about your breathing and any symptoms you may be experiencing. This should take about 10 minutes. After radiation therapy is complete, some of the monthly questionnaires will be completed by the data coordinator using telephone interviews.

Length of Study:

Your participation in this study will be over after you complete the last breath testing session.

This is an investigational study. The nitric oxide breath analyzer used in this study is FDA approved and commercially available for measuring breathed out nitric oxide levels in patients with asthma. Its use to predict lung inflammation caused by radiation therapy is investigational.

Up to 150 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will sign consent for the study.
2. Patients with pathologic diagnosis of esophagus or lung cancer.
3. Patient plans to receive radiation treatment at MD Anderson.
4. Patient will receive >/= 5 weeks of thoracic radiotherapy.
5. Patients >/= 18 years of age.

Exclusion Criteria:

1. Patients who have asthma.
2. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide) throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung and esphageal cancer patients receiving radiation therapy, at UT MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Ratio Between Weekly and Baseline Nitric Oxide (NO) Measurements | Weekly starting prior to start of radiation therapy to follow-up visits for 6 months.
  Ratio between weekly and baseline nitric oxide measurements in participants receiving thoracic radiation therapy. Exhaled nitric oxide measured in triplicate on a weekly basis during radiotherapy and on each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Guerrero, MD, PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Website — http://www.mdanderson.org